CLINICAL TRIAL: NCT01886534
Title: A Randomized Controlled Trial of Enhanced Caregiver Support Versus Usual Care for Managing Older Heart Failure Patients at Hospital Discharge
Brief Title: Caregiver Enhanced Assistance and Support for the Elderly Heart Failure Patient at Hospital Discharge (CEASE-HF)
Acronym: CEASE-HF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Catherine Demers, Associate Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11-638
Record Dates: First submitted 2013-06-21; First posted 2013-06-26 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Heart Failure
Keywords: Heart failure; Heart diseases; Cardiovascular diseases; Health information technology; Disease management; Patient care management; Self care; Informal caregiver; Care partner; Peer support; Transitional care; Patient education; Teach-back; Clinical decision aid
MeSH Terms: conditions — Heart Failure; Heart Diseases; Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Enhanced Caregiver Support with Caregiver (Experimental): * Standardized Heart Failure Discharge Summary to Primary Care Physicians©
  * Standardized education sessions
  * Heart Failure Diuretic Decision Support Tool for Patient Self Management©
  * Digital talking scale
  Interventions: Other: Standardized Heart Failure Discharge Summary to Primary Care Physicians©; Behavioral: Standardized education sessions; Other: Heart Failure Diuretic Decision Support Tool for Patient Self Management©; Other: Digital talking scale; Other: Usual care
- Usual Care with Caregiver (Other): * Usual care
  Interventions: Other: Usual care
- Enhanced Support without Caregiver (Experimental): * Standardized Heart Failure Discharge Summary to Primary Care Physicians©
  * Standardized education sessions
  * Heart Failure Diuretic Decision Support Tool for Patient Self Management©
  * Digital talking scale
  Interventions: Other: Standardized Heart Failure Discharge Summary to Primary Care Physicians©; Behavioral: Standardized education sessions; Other: Heart Failure Diuretic Decision Support Tool for Patient Self Management©; Other: Digital talking scale; Other: Usual care
- Usual Care without Caregiver (Other): * Usual Care
  Interventions: Other: Usual care

INTERVENTIONS:
Other: Standardized Heart Failure Discharge Summary to Primary Care Physicians© — At hospital discharge, in addition to usual care, the Study Nurse will fax an introduction letter and a 1-page comprehensive Standardized Heart Failure Discharge Summary to Primary Care Physicians© integrating Canadian Cardiovascular Society HF guideline recommendations to the patient's family physician.
  Arms: Enhanced Caregiver Support with Caregiver; Enhanced Support without Caregiver
Behavioral: Standardized education sessions — Following baseline data collection, and prior to hospital discharge or within 72 hours of discharge, all patient/caregiver dyads in the intervention group will receive a 45-60-minute standardized education session with the study nurse according to individualized patient learning needs, aimed to ensure similar baseline level of heart failure self-care knowledge. Verbal (teach-back) and written information from the Trial of Education And Compliance in Heart dysfunction (TEACH) RCT will be provided to all patient/caregiver dyads. Information regarding self-care such as dietary restrictions, exercise guidelines, weight and symptom monitoring (shortness of breath, swelling of the ankles) included in the education package will be reviewed. The teaching sessions will occur at 1 week, 2 weeks, 1 month and 2 months post-discharge.
  Arms: Enhanced Caregiver Support with Caregiver; Enhanced Support without Caregiver
Other: Heart Failure Diuretic Decision Support Tool for Patient Self Management© — Each patient/caregiver dyad will be provided a paper-based Heart Failure Diuretic Decision Support Tool for Patient Self Management© at hospital discharge assisting in the titration of their oral furosemide. The purpose of this tool will be to assist the patient/caregiver in keeping track of signs and symptoms of worsening heart failure. The family physician will also be provided an access to similar decision support tool for management of clinical deterioration.
  Arms: Enhanced Caregiver Support with Caregiver; Enhanced Support without Caregiver
Other: Digital talking scale — Prior to hospital discharge, the patient/caregiver dyad will be provided a digital, talking scale to measure their weight in their home setting.
  Arms: Enhanced Caregiver Support with Caregiver; Enhanced Support without Caregiver
Other: Usual care — Patients allocated to the usual care group will receive the hospital-approved heart failure management booklet which meets evidence-based requirements for outpatient heart failure management. Patients will meet with the hospital HF nurse-clinician (standard at this institution) to review heart failure symptoms and signs, diet and exercise recommendations. They will also meet with the ward pharmacist prior to hospital discharge to review medications and side effects. Referral to the HF clinic and any HF initiative will be left to the discretion of the most responsible physician.

SUMMARY:
Close to ninety percent of older heart failure (HF) patients have some cognitive deficits at hospital discharge which may impact their ability to make effective decisions about their healthcare. However, informal care partners (CPs) may assist in managing HF when provided with appropriate education and support. The goal of this randomized clinical trial (RCT) is to evaluate an intervention which will provide 1) additional teaching on management of HF to the patient and CP following hospital discharge, 2) improved communication with the family physician, 3) a HF decision support tool for oral diuretic management, and 4) a digital talking scale. The investigators believe this intervention will improve outcomes and be cost saving.

The investigators hypothesize that enhanced education and support for the CPs to assist older HF patients following hospital discharge, combined with improved communication with family physicians, contact with a HF nurse, and simple decision support tools, will lead to earlier recognition of clinical deterioration, and improved patient outcomes. Innovative and cost-effective approaches to manage HF patients following hospital discharge are urgently needed in Canada.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Heart Failure (with preserved or impaired left ventricular systolic dysfunction) confirmed with the Boston Criteria >= 5 points
* 60 years of age or older

Exclusion Criteria:

* Residence in, or planned discharge to a long-term care facility (LTC)
* Life expectancy less than 3 months
* Patient transferred to Geriatric Rehabilitation unit
* No caregiver
* Residence is more than a 30 minute rive from hospital of discharge
* Patient refused to participate
* Caregiver refused to participate
* Patient referred for CV surgery prior to hospital discharge
* Patient on IV Lasix at or bumetamide at hospital discharge
* Not on PO Lasix at hospital discharge
* Patient currently on dialysis
* Caregiver unavailable during daytime hours
* Caregiver has disability, serious mental illness or cognitive dysfunction
* Patient discharged early
* Patient enrolled in another randomized controlled trial
* Patient expired
* Patient and caregiver unable to speak and read English (Patient may be enrolled if nurse can converse minimally with patient and caregiver. S-TOFHLA will not be done for reading comprehension and questionnaires will be administered orally.)
* Severe aortic stenosis or severe mitral stenosis

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2012-09; Primary Completion 2014-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Patient self care | 3 months
  Self-Care Heart Failure Index (SCHFI) for patients and caregivers

SECONDARY OUTCOMES:
Death | 3 months
  Deaths (due to cardiac and non-cardiac causes) during 3 months after hospital discharge
Heart failure readmission | 3 months
  Heart failure readmission (>= 24 hour hospital stay including the time spent in the emergency room with clinical evidence of heart failure) during 3 months after hospital discharge
Emergency room heart failure visits | 3 months
  Emergency room heart failure visits (< 24 hour hospital stay) during 3 months after hospital discharge
Perceived caregiver burden | 3 months
  Modified Oberst Caregiver Burden Scale (CBS)
Heart failure knowledge acquisition | 3 months
  Knowledge Acquisition Questionnaire (KAQ) for patients and caregivers
Medication adherence | 3 months
  Medication Possession Ratio (MPR)
Referral to heart failure clinic or to long-term care | 3 months
Health beliefs | 3 months
  Health Beliefs Questionnaire (HBQ) for patients and caregivers
Depression | 3 months
  Geriatric Depression Scale 8 (GDS-8) for the patient

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Demers, MD, MSc, FRCPC, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada